CLINICAL TRIAL: NCT00241423
Title: Effect of Exenatide on 24-Hour Blood Glucose Profile Compared With Placebo in Patients With Type 2 Diabetes Using Metformin or Metformin Plus a Thiazolidinedione
Brief Title: Effect of Exenatide on 24-Hour Blood Glucose Profile Compared With Placebo in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-US-GWAW
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide; diabetes; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Exenatide and the subject's current oral antidiabetic agent regimen
  Interventions: Drug: exenatide
- Placebo (Placebo Comparator): Placebo and the subject's current oral antidiabetic agent regimen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg twice a day for one week; then 10 mcg twice a day for one week
  Other Names: Byetta; AC2993; synthetic enxendin-4
  Arms: Exenatide
Drug: Placebo — subcutaneous injection, equivalent volume to 5 mcg exenatide twice a day for one week; then equivalent volume to 10 mcg exenatide twice a day for one week
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that in patients with type 2 diabetes, the addition of exenatide will result in lower time-averaged serum glucose during a 24-hour period, compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject has an HbA1c between 7.0% and 10.0%, inclusive.
* Subject has a body mass index (BMI) >25 kg/m^2 and <50 kg/m^2.
* Subject is on a stable dose of metformin or metformin plus a thiazolidinedione.

Exclusion Criteria:

* Subject has been treated with any of the following medications: *exogenous insulin for more than 1 week within 3 months of screening, *sulfonylureas or meglitinides within 2 months of screening, *alpha-glucosidase inhibitors within 2 months of screening, *pramlintide acetate injection within 2 months of screening.
* Subject has received exenatide, GLP-1 analogs, DPP-IV inhibitors, or has participated in this study previously.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Time-averaged serum glucose during a 24-hour period | Every half-hour to hour for 24 hours
  Time-averaged serum glucose during a 24-hour period

SECONDARY OUTCOMES:
To compare the effects of exenatide and placebo on serum glucose | Each half-hour to 2 hours for 24 hours
  To compare the effects of exenatide and placebo on serum glucose measured as averaged daytime glucose, averaged nighttime glucose, time-averaged postprandial glucose 2 hours after each meal, time-averaged postprandial glucose 4 hours after each meal, 2-hour postprandial glucose averaged across morning and evening meals, and averaged across the three meals, and fluctuation evaluations

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Research Site, Washington D.C., District of Columbia
  - Research Site, San Antonio, Texas

REFERENCES:
- [Derived] Brodows RG, Qu Y, Johns D, Kim D, Holcombe JH. Quantifying the effect of exenatide and insulin glargine on postprandial glucose excursions in patients with type 2 diabetes. Curr Med Res Opin. 2008 May;24(5):1395-7. doi: 10.1185/030079908x297268. Epub 2008 Apr 3. PMID 18394265